CLINICAL TRIAL: NCT03841942
Title: Comparison of Trough Level-based Spacing and Clinical-based Spacing of Infliximab Infusions in Patients With Inflammatory Bowel Disease in Deep Remission; A Prospective, Multicenter, Open-label, Randomized, Controlled Study
Brief Title: Comparison of Trough Level- and Clinical-based Spacing of Infliximab Infusions in Patients With IBD in Deep Remission
Acronym: SPACIFIX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty of inclusion
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL18_0024 7596
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clinically-based spacing (Other): All patients (as there are free from symptoms) after inclusion will have a spacing of their infliximab infusion interval which will be maintained until the end of the study.
  Interventions: Other: clinically-based spacing strategy
- Trough level-based spacing (Other): Only patients with a baseline infliximab trough level ≥ 7 ug/ml will have a spacing of their infliximab infusion interval which will be maintained until the end of the study. Patients with a baseline infliximab trough level < 7 ug/ml will keep their baseline infliximab infusion interval until the end of the study.
  Interventions: Other: Trough level-based strategy

INTERVENTIONS:
Other: clinically-based spacing strategy — All patients (as there are free from symptoms) will have a first step of a 2 weeks spacing of their infliximab infusion interval. Then, at the next infliximab infusion, if clinical remission is maintained (CDAI < 150 for CD, Partial Mayo score < 3 for UC), patients will have a second step of a 2 weeks infliximab infusion spacing which will be maintained until the end of the study.
  Arms: clinically-based spacing
Other: Trough level-based strategy — patients will have at inclusion a determination of the infliximab trough level. According to this dosage, only patients with a trough level ≥ 7 µg/ml will have a first step of a 2 weeks spacing of their infliximab infusion interval. Then, at the next infliximab infusion, if clinical remission (CDAI < 150 for CD, Partial Mayo score < 3 for UC) is maintained and if infliximab trough level is still ≥ 7 ug/ml, patients will have a second step of 2 weeks infliximab spacing until the end of the study.
  Patients with a baseline infliximab trough level < 7 ug/ml will keep their baseline infliximab infusion interval until the end of the study.
  Arms: Trough level-based spacing

SUMMARY:
Comparison of trough level-based spacing and clinical-based spacing of infliximab infusions in patients with inflammatory bowel disease in deep remission A prospective, multicenter, open-label, randomized, controlled Study

DETAILED DESCRIPTION:
Infliximab (IFX) is common treatment for refractory inflammatory bowel disease (IBD) (5 mg/kg/8 weeks in maintenance). A large majority of IBD patients treated with IFX are currently in long-term clinical remission under maintenance IFX monotherapy or cotherapy with azathioprine or methotrexate. There is no recommendation on optimal duration of anti-TNF therapy once it is started. A key question is to know if the treatment could be stopped/decreased without clinical relapse. Anti-TNF therapy is also a major burden in health care costs in France. Identifying an optimal duration of anti-TNF therapy and criteria for stopping/decreasing could help in lowering these therapies cost without altering disease control. Prospective studies have investigated the withdrawal of IFX in IBD patients showing 50% of clinical relapse at 1 year in patient in clinical remission, 30% in patients in deep remission.

Another alternative to deescalate anti-TNF treatment would be to increase the infusion interval without stopping the drug. Indeed, this infusion interval spacing is strongly requested by patients who seek an improvement in their quality of life. This empirical spacing corresponded to an increase of the infusion interval to 10 weeks then to 12 weeks maximum in patients with persistent clinical remission. In France and in Europe, even if there is no recommendation about infliximab de-escalation and increase of the infusion interval, many physicians have already performed empirically an infliximab infusion interval spacing in IBD patients in longstanding remission while on infliximab maintenance therapy. This empirical infusion interval increase in patients in clinical remission leads to a clinical relapse in 30% of these patients with a median delay of 12.6 months (IQR: 10.4- 18.4) (Dufour et al. UEGW 2017).

Since the last ten years, it was demonstrated that the serum level of infliximab measured just before the last infliximab infusion (defined as a trough level) is correlated to the clinical activity of the disease1. A serum IFX trough level between 3 and 7 ug/ml has been identified as therapeutic with more clinical relapse in patients with IFX < 3 ug/ml and safe dose reduction in patients with IFX trough level > 7 ug/ml.

Thus, we hypothesized that using the determination of serum infliximab trough level could decrease the risk of clinical relapse observed in IBD patients who underwent an empirical infliximab infusion interval spacing (approximatively 30% of the cases). Indeed, in an infliximab trough level-based spacing strategy, only patients with a supratherapeutic (>7ug/ml) infliximab trough level would have a spacing of infliximab infusion.

The aim of our study is to compare an IFX infusion interval spacing strategy based on IFX trough level with an IFX infusion interval spacing strategy based on clinical evaluation for maintaining clinical and biological remission in IBD patients in deep remission.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years

  * Patients with a diagnosis of Crohn's disease or ulcerative colitis according to clinical, biological, morphological and endoscopic criteria defined by the ECCO guidelines22, 23
  * Patients in deep remission since at least 6 months17:

    * CDAI < 150 for CD, Partial Mayo score < 3 for UC
    * CRP (C reactive protein) < 10 mg/l
    * CDEIS < 6 (<3 in each segment) for CD, Mayo endoscopic subscore of 0 or 1 for UC
    * For CD patients with small bowel disease: No ulceration on MRI, only asymptomatic fibrotic stenosis without inflammation and retro dilatation. No ulceration on wireless capsule endoscopy if feasible
    * For patients with perianal disease: No active draining fistula, or perianal abscess on clinical exam and MRI
  * Treatment with infliximab at stable dose (5mg/kg) with a stable interval for at least 4 months
  * Infliximab trough level > 3 ug/ml
  * No change in other IBD therapies in the past 4 months
  * Signed informed consent form
  * Subjects must be able to attend all scheduled visits and to comply with all trial procedures
  * Subjects must be covered by public health insurance

Exclusion Criteria:

* Subject unable to read or/and write

  * Planned longer stay outside the region that prevents compliance with the visit plan
  * Subject who are in a dependency or employment with the sponsor or the investigator
  * Participation in another clinical trial or administration of an unapproved drug within the last 4 weeks before the screening date
  * Previous withdrawal or spacing over 8 weeks of infliximab therapy
  * Infliximab therapy at 10 mg/kg
  * Patients who have presented a severe acute or delayed reaction to infliximab.
  * Active perianal/abdominal fistulae at time of inclusion, defined by active drainage
  * Patients with ostomy or ileoanal pouch
  * Pregnancy or planned pregnancy during the study
  * Inability to follow study procedures as judged by the investigator
  * Steroid use ≤3 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Rate of loss of clinical remission | 12 months
  mucosal Healing
Rate of loss of biological remission | 12 months
  antidrug antibodies with detectable IFX trough levels

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Pineton de Chambrun, Principal Investigator — CHU of Montpellier
Locations (16):
- France (16):
  - Amiens University Hospital, Amiens
  - Besançon University Hospital, Besançon
  - Bordeaux University Hospital, Bordeaux
  - Caen University Hospital, Caen
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - Lille University Hospital, Lille
  - Pineton de Chambrun, Montpellier
  - CHRU Nancy - Hôpitaux de Brabois, Nancy
  - Nantes University Hospital, Nantes
  - Nice University Hospital, Nice
  - Nîmes University Hospital, Nîmes
  - APHP Beaujon Hospital, Paris
  - APHP Paris Cochin, Paris
  - Rennes University Hospital, Rennes
  - Saint Etienne University Hospital, Saint-Etienne
  - Toulouse University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No